CLINICAL TRIAL: NCT03786926
Title: A Phase 1, Open-Label Study to Evaluate the Safety, Tolerability, Pharmacokinetics and Preliminary Efficacy of HMPL-689 in Patients With Relapsed or Refractory Lymphoma
Brief Title: Trial to Evaluate the Safety and Pharmacokinetics of HMPL-689 in Patients With Lymphomas
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: 2018-689-00US1 has been halted by HUTCHMED based on strategic evaluation of the clinical development of HMPL-689 in the United States, Europe, and Australia.
Sponsor: Hutchmed (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2018-689-00US1
Record Dates: First submitted 2018-12-18; First posted 2018-12-26 (Actual); Results first posted 2025-06-26 (Actual); Last update posted 2025-06-26 (Actual); Status verified 2025-06

CONDITIONS: Lymphoma
Keywords: CLL; SLL; FL; MZL; LPL; WM; MCL; PTCL; CBCL
MeSH Terms: conditions — Lymphoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (Experimental): All patients take HMPL-689 taken daily
  Interventions: Drug: HMPL-689

INTERVENTIONS:
Drug: HMPL-689 — HMPL-689 is a PI3Kδ inhibitor

SUMMARY:
An open-label, dose escalation and expansion clinical trial to evaluate the safety, tolerability and PK of HMPL-689 in patients with relapsed or refractory lymphomas

DETAILED DESCRIPTION:
This is a Phase 1, open-label, multicenter study of HMPL-689 administered orally to patients with relapsed or refractory lymphoma.

HMPL-689 is a selective and potent small molecule inhibitor targeting the isoform phosphoinositide 3'-kinase delta (PI3Kδ), a key component in the B-cell receptor signaling pathway

This study will consist of a dose escalation stage (Stage 1) and a dose expansion stage (Stage 2).

Dose Escalation Stage (Stage 1):

This stage will end when any of the following criteria is met:

* The dose level 1 demonstrates an excessive toxicity, ie, 3 dose limiting toxicities (DLTs) are observed out of the first 3 patients at dose level 1.
* The maximum sample size is reached.
* The MTD and/or RP2D is confirmed.

Dose Expansion Stage (Stage 2):

To further characterize the safety and explore the preliminary anti-tumor activity of HMPL-689 at RP2D, patients with B cell lymphoma will be enrolled in the dose expansion stage.

ELIGIBILITY:
Inclusion Criteria:

1. (ECOG) performance status of 0 or 1;
2. Histologically confirmed lymphoma (tumor types are restricted to CLL/SLL, FL (grade 1-3a), MCL, MZL, LPL/WM, PTCL or CBCL);
3. Patients with relapsed or refractory NHL for whom:

   * Standard of care treatment options no longer exist (Stage 1 only);
   * Standard of care treatment options no longer exist with the exception of PI3K-delta inhibitors (Stage 2 only);
4. Expected survival of more than 24 weeks.

Exclusion Criteria:

Patients who meet any of the following criteria will be excluded from study entry:

1. Primary central nervous system (CNS) lymphoma;
2. Any of the following laboratory abnormalities Absolute neutrophil count; <1.0×10^9/L, Hemoglobin <80 g/L Platelets <50 ×10^9/L
3. Inadequate organ function, defined by the following:

   * Total bilirubin ≥1.5 times the upper limit of normal (× ULN);
   * AST or ALT > 2.5 × ULN;
   * Estimated creatinine clearance (CrCl) per Cockcroft-Gault;
   * Dose Escalation stage of trial (Stage 1) - CrCl < 40 mL/min;
   * Dose Expansion stage of trial (Stage 2) - CrCl <30 mL/min;
4. International normalized ratio (INR) > 1.5 × ULN, activated partial thromboplastin time (aPTT) > 1.5 × ULN;
5. Serum amylase or lipase > ULN at screening or known medical history of serum amylase or lipase > ULN;
6. Patients with presence of second primary malignant tumors within the last 2 years;
7. Clinically significant history of liver disease;
8. Prior treatment with any PI3Kδ inhibitors;
9. Any prior use of the following: cancer therapy within 3 weeks of study treatment, GCSF within 7 days of screening, steroid therapy or targeted anti-neoplastic intent within 7 days of treatment, any use of strong CYP3A4 inducers within 2 weeks prior to initiation of study treatment, prior autologous transplant within 6 months of study treatment, prior allogenic stem cell transplant within 6 months of study treatment;
10. Clinically significant active infection or interstitial lung diseases (including drug induced pneumonitis);
11. Major surgical procedure within 4 weeks prior to initiation of study treatment;
12. Adverse events from prior anti-neoplastic therapy that have not resolved to Grade less than or equal to 1, except for alopecia;
13. New York Heart Association (NYHA) Class II or greater congestive heart failure;
14. Congenital long QT syndrome or QTc >470 msec;
15. Currently use medication known to cause QT prolongation or torsades de pointes;
16. History of myocardial infarction or unstable angina within 6 months prior to initiation of study treatment;
17. History of stroke or transient ischemic attack within 6 months prior to initiation of study treatment;
18. Inability to take oral medication, prior surgical procedures affecting absorption, or active peptic ulcer disease;
19. History of inflammatory bowel disease (e.g., Crohn's disease or ulcerative colitis);
20. Patients with ongoing chronic gastrointestinal diseases;
21. Any other diseases, metabolic dysfunction, physical examination finding, or clinical laboratory finding that, in the investigator's opinion, gives reasonable suspicion of a disease or condition that contraindicates the use of an investigational drug or that may affect the interpretation of the results or renders the patient at high risk from treatment complications.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2019-08-26 (Actual); Primary Completion 2024-06-26 (Actual); Study Completion 2024-06-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Claudia Huang, Study Director — Hutchmed Limited; Nilanjan Ghosh, MD, Principal Investigator — Atrium Health Levine Cancer Institute; Jonathan B Cohen, MD, Principal Investigator — Emory Winship Cancer Institute
Locations (27):
- United States (10):
  - Innovative Clinical Research Institute, Anaheim, California
  - Pacific Cancer Medical Center, Anaheim, California
  - Ventura County Hematology-Oncology Specialists, Oxnard, California
  - Winship Cancer Institute of Emory University, Atlanta, Georgia
  - Clinical Research Alliance, Inc, Westbury, New York
  - Levine Cancer Institute- Atrium Health, Charlotte, North Carolina
  - Baylor Scott and White Research Institute, Dallas, Texas
  - Renovatio Clinical, Houston, Texas
  - University of Texas Health Science Center at San Antonio, San Antonio, Texas
  - Medical Oncology Associates, P.S., Spokane, Washington
- Finland (2):
  - Helsingin yliopistollinen keskussairaala, Helsinki
  - Tampereen yliopistollinen sairaala, Tampere
- France (3):
  - Hopital Henri Mondor, Créteil, Val De Marne
  - CHU de Nantes - Hotel Dieu, Nantes
  - CHU de Bordeaux - Hôpital Haut-Lévêque, Pessac
- Italy (2):
  - Azienda Ospedaliera Universitaria Policlinico Sant'Orsola Malpighi IRCCS, Bologna
  - Ospedale San Raffaele, Milan
- Poland (5):
  - KO-MED Centra Kliniczne, Biała Podlaska
  - Uniwersyteckie Centrum Kliniczne, Gdansk
  - BioResearch Group Sp. Z. o. o., Krakow
  - NASZ LEKARZ Osrodek Badan Klinicznych, Torun
  - Uniwersytecki Szpital Kliniczny im. Jana Mikulicza Radeckiego, Wroclaw
- Spain (5):
  - ICO Badalona - Hospital Universitari Germans Trias i Pujol, Barcelona
  - ICO l'Hospitalet - Hospital Duran i Reynals, Barcelona
  - Fundacion Jimenez Diaz, Madrid
  - Hospital Universitario Virgen del Rocio, Seville
  - Hospital Universitario Virgen Macarena, Seville

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This Phase 1, 2-part, open-label study was conducted in patients with relapsed, refractory, or resistant lymphoma.
Pre-assignment Details: The study consisted of a dose escalation stage (stage 1) and a dose expansion stage (stage 2). A total of 23 patients in dose escalation stage and 30 patients in dose expansion stage were enrolled in this study. The study was terminated based on strategic evaluation of the clinical development of HMPL-689 in the United States, Europe, and Australia with no safety concerns.
Groups:
- Dose Escalation Stage: HMPL-689 5 mg QD: Patients received HMPL-689 5 milligram (mg) once daily (QD) orally for continuous 28-day treatment cycles until disease progression (PD), death, intolerable toxicity, investigator's assessment of no benefit from the study treatment, withdrawal from the study, or the end of study, whichever occurred first.
- Dose Escalation Stage: HMPL-689 10 mg QD: Patients received HMPL-689 10 mg QD orally for continuous 28-day treatment cycles until PD, death, intolerable toxicity, investigator's assessment of no benefit from the study treatment, withdrawal from the study, or the end of study, whichever occurred first.
- Dose Escalation Stage: HMPL-689 15 mg QD: Patients received HMPL-689 15 mg QD orally for continuous 28-day treatment cycles until PD, death, intolerable toxicity, investigator's assessment of no benefit from the study treatment, withdrawal from the study, or the end of study, whichever occurred first.
- Dose Escalation Stage: HMPL-689 20 mg QD: Patients received HMPL-689 20 mg QD orally for continuous 28-day treatment cycles until PD, death, intolerable toxicity, investigator's assessment of no benefit from the study treatment, withdrawal from the study, or the end of study, whichever occurred first.
- Dose Escalation Stage: HMPL-689 25 mg QD: Patients received HMPL-689 25 mg QD orally for continuous 28-day treatment cycles until PD, death, intolerable toxicity, investigator's assessment of no benefit from the study treatment, withdrawal from the study, or the end of study, whichever occurred first.
- Dose Escalation Stage: HMPL-689 30 mg QD: Patients received HMPL-689 30 mg QD orally for continuous 28-day treatment cycles until PD, death, intolerable toxicity, investigator's assessment of no benefit from the study treatment, withdrawal from the study, or the end of study, whichever occurred first.
- Dose Expansion Stage: CLL/SLL: Patients with chronic lymphocytic leukemia (CLL)/small lymphocytic lymphoma (SLL) received HMPL-689 at recommended phase 2 dose (RP2D), that is, 30 mg QD orally for continuous 28-day treatment cycles until PD, death, intolerable toxicity, investigator's assessment of no benefit from the study treatment, withdrawal from the study, or the end of study, whichever occurred first.
- Dose Expansion Stage: FL: Patients with follicular lymphoma (FL) received HMPL-689 at RP2D, that is, 30 mg QD orally for continuous 28-day treatment cycles until PD, death, intolerable toxicity, investigator's assessment of no benefit from the study treatment, withdrawal from the study, or the end of study, whichever occurred first.
- Dose Expansion Stage: MZL: Patient with marginal zone lymphoma (MZL) received HMPL-689 at RP2D, that is, 30 mg QD orally for continuous 28-day treatment cycles until PD, death, intolerable toxicity, investigator's assessment of no benefit from the study treatment, withdrawal from the study, or the end of study, whichever occurred first.
- Dose Expansion Stage: LPL/WM: Patients with lymphoplasmacytic lymphoma/Waldenström's macroglobulinemia (LPL/WM) received HMPL-689 at RP2D, that is, 30 mg QD orally for continuous 28-day treatment cycles until PD, death, intolerable toxicity, investigator's assessment of no benefit from the study treatment, withdrawal from the study, or the end of study, whichever occurred first.
- Dose Expansion Stage: MCL: Patients with mantle cell lymphoma (MCL) received HMPL-689 at RP2D, that is, 30 mg QD orally for continuous 28-day treatment cycles until PD, death, intolerable toxicity, investigator's assessment of no benefit from the study treatment, withdrawal from the study, or the end of study, whichever occurred first.
Period: Overall Study
Arm/Group | Dose Escalation Stage: HMPL-689 5 mg QD | Dose Escalation Stage: HMPL-689 10 mg QD | Dose Escalation Stage: HMPL-689 15 mg QD | Dose Escalation Stage: HMPL-689 20 mg QD | Dose Escalation Stage: HMPL-689 25 mg QD | Dose Escalation Stage: HMPL-689 30 mg QD | Dose Expansion Stage: CLL/SLL | Dose Expansion Stage: FL | Dose Expansion Stage: MZL | Dose Expansion Stage: LPL/WM | Dose Expansion Stage: MCL
Started | 3 | 3 | 5 | 3 | 6 | 3 | 3 | 13 | 6 | 3 | 5
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 3 | 3 | 5 | 3 | 6 | 3 | 3 | 13 | 6 | 3 | 5
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 1
Not completed — Progressive disease | 3 | 0 | 3 | 1 | 2 | 2 | 1 | 6 | 1 | 1 | 1
Not completed — Death | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2
Not completed — Physician Decision | 0 | 1 | 0 | 1 | 2 | 0 | 0 | 2 | 1 | 1 | 0
Not completed — Withdrawal by Subject | 0 | 1 | 1 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 1
Not completed — Study terminated by Sponsor | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 4 | 0 | 0 | 0
Not completed — Anti-neoplasm treatment | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Other | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 2 | 0 | 0

BASELINE CHARACTERISTICS:
Population: The Full Analysis Set (FAS) included all patients who received at least 1 dose of HMPL-689.
Groups:
- Dose Escalation Stage: HMPL-689 5 mg QD: Patients received HMPL-689 5 mg QD orally for continuous 28-day treatment cycles until PD, death, intolerable toxicity, investigator's assessment of no benefit from the study treatment, withdrawal from the study, or the end of study, whichever occurred first.
- Dose Expansion Stage: CLL/SLL: Patients with CLL/SLL received HMPL-689 at RP2D, that is, 30 mg QD orally for continuous 28-day treatment cycles until PD, death, intolerable toxicity, investigator's assessment of no benefit from the study treatment, withdrawal from the study, or the end of study, whichever occurred first.
- Dose Expansion Stage: FL: Patients with FL received HMPL-689 at RP2D, that is, 30 mg QD orally for continuous 28-day treatment cycles until PD, death, intolerable toxicity, investigator's assessment of no benefit from the study treatment, withdrawal from the study, or the end of study, whichever occurred first.
- Dose Expansion Stage: MZL: Patient with MZL received HMPL-689 at RP2D, that is, 30 mg QD orally for continuous 28-day treatment cycles until PD, death, intolerable toxicity, investigator's assessment of no benefit from the study treatment, withdrawal from the study, or the end of study, whichever occurred first.
- Dose Expansion Stage: LPL/WM: Patients with LPL/WM received HMPL-689 at RP2D, that is, 30 mg QD orally for continuous 28-day treatment cycles until PD, death, intolerable toxicity, investigator's assessment of no benefit from the study treatment, withdrawal from the study, or the end of study, whichever occurred first.
- Dose Expansion Stage: MCL: Patients with MCL received HMPL-689 at RP2D, that is, 30 mg QD orally for continuous 28-day treatment cycles until PD, death, intolerable toxicity, investigator's assessment of no benefit from the study treatment, withdrawal from the study, or the end of study, whichever occurred first.
- Total: Total of all reporting groups
Arm/Group | Dose Escalation Stage: HMPL-689 5 mg QD | Dose Escalation Stage: HMPL-689 10 mg QD | Dose Escalation Stage: HMPL-689 15 mg QD | Dose Escalation Stage: HMPL-689 20 mg QD | Dose Escalation Stage: HMPL-689 25 mg QD | Dose Escalation Stage: HMPL-689 30 mg QD | Dose Expansion Stage: CLL/SLL | Dose Expansion Stage: FL | Dose Expansion Stage: MZL | Dose Expansion Stage: LPL/WM | Dose Expansion Stage: MCL | Total
Number analyzed (Participants) | 3 | 3 | 5 | 3 | 6 | 3 | 3 | 13 | 6 | 3 | 5 | 53
Age, Continuous [Mean (Standard Deviation); unit: years] | 69.7 (6.51) | 70.7 (13.05) | 64.8 (17.18) | 67.7 (3.51) | 63.8 (7.68) | 59.0 (17.69) | 65.7 (5.03) | 61.7 (10.16) | 72.3 (9.56) | 63.7 (4.16) | 75.8 (8.23) | 66.2 (10.63)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 2 | 0 | 0 | 3 | 1 | 2 | 9 | 1 | 1 | 1 | 21
  Male | 2 | 1 | 5 | 3 | 3 | 2 | 1 | 4 | 5 | 2 | 4 | 32
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 3 | 3 | 5 | 3 | 5 | 3 | 3 | 13 | 6 | 3 | 5 | 52
  Other | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 2 | 0 | 0 | 1 | 0 | 0 | 3 | 1 | 0 | 2 | 9
  Not Hispanic or Latino | 3 | 1 | 5 | 3 | 5 | 3 | 3 | 10 | 4 | 3 | 3 | 43
  Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Dose Escalation Stage: Number of Patients With Dose-Limiting Toxicities (DLTs)
Description: A DLT was defined as the occurrence of any of the following treatment-emergent adverse events (TEAEs) during the DLT assessment window, unless equivocally due to underlying malignancy or an extraneous cause. AEs were graded using National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version 5.0: non-hematologic toxicity: all non-hematologic TEAEs of grade 3 or greater with the exception of grade 3 nausea or vomiting that could be controlled by supportive therapy; hematologic toxicity: grade 4 neutropenia >5 days, grade 4 thrombocytopenia or grade 3 thrombocytopenia with bleeding event or requiring platelet transfusion, grade >=3 febrile neutropenia (defined as absolute neutrophil count [ANC] <1000/cubic millimeter {mm^3} with a single temperature >38.3 degree Celsius [°C] or a sustained temperature of >=38°C for more than 1 hour), grade 4 anemia not explained by underlying disease; any TEAE that required a dose delay of >=15 days; any case of Hy's Law.
Time Frame: From the first dose of study drug (Day 1) up to Day 28 of Cycle 1 (each cycle is 28 days)
Population: The DLT evaluable analysis set (DEAS) was defined as all patients enrolled in the dose escalation stage of the study who were evaluable for DLT assessment. A patient was DLT evaluable if: had received at least 75% of the assigned dose of study drug during the DLT assessment window or had not completed the DLT assessment period due to a DLT.
Measure: Count of Participants; unit: Participants
Arm/Group | Dose Escalation Stage: HMPL-689 5 mg QD | Dose Escalation Stage: HMPL-689 10 mg QD | Dose Escalation Stage: HMPL-689 15 mg QD | Dose Escalation Stage: HMPL-689 20 mg QD | Dose Escalation Stage: HMPL-689 25 mg QD | Dose Escalation Stage: HMPL-689 30 mg QD
Number analyzed (Participants) | 3 | 3 | 5 | 3 | 6 | 3
Participants | 0 | 0 | 1 | 0 | 1 | 0

2. Primary Outcome: Dose Escalation Stage: Number of Patients With Treatment-Emergent Adverse Events (TEAEs), Treatment Related Treatment-Emergent Adverse Events (TRAEs), Treatment-Emergent Serious Adverse Events (TESAEs) and Treatment Related Serious Adverse Events (TRSAEs)
Description: An AE was any untoward medical occurrence in a clinical investigation patient administered a study drug, regardless of causal attribution. An SAE was an AE that resulted in any of the following: was fatal, was life threatening, required or prolonged inpatient hospitalization, resulted in persistent or significant disability/incapacity, was a congenital anomaly/birth defect in a neonate/infant born to a female patient or female partner of a male patient exposed to the study drug, or was considered a significant medical event by the investigator. TEAEs were defined as AEs with onset date on or after the first dose of study drug and no later than 30 days after the date of last study drug administration or start of a new study drug of anti-neoplasm therapy, whichever was earlier. Treatment related AEs and SAEs were defined as AEs and SAEs collected later than 30 days after the last study drug date or start of a new study drug of anti-neoplasm therapy.
Time Frame: From the first dose of study drug (Day 1) up to 30 days after the last dose of study drug, approximately 34 months
Population: The FAS included all patients who received at least 1 dose of HMPL-689.
Measure: Count of Participants; unit: Participants
Arm/Group | Dose Escalation Stage: HMPL-689 5 mg QD | Dose Escalation Stage: HMPL-689 10 mg QD | Dose Escalation Stage: HMPL-689 15 mg QD | Dose Escalation Stage: HMPL-689 20 mg QD | Dose Escalation Stage: HMPL-689 25 mg QD | Dose Escalation Stage: HMPL-689 30 mg QD
Number analyzed (Participants) | 3 | 3 | 5 | 3 | 6 | 3
Participants
  Any TEAE | 3 | 3 | 5 | 3 | 6 | 3
  Any TRAE | 1 | 3 | 4 | 3 | 6 | 3
  Any TESAE | 0 | 2 | 2 | 3 | 2 | 1
  Any TRSAE | 0 | 0 | 1 | 2 | 2 | 0

3. Primary Outcome: Dose Expansion Stage: Number of Patients With Treatment-Emergent Adverse Events and Treatment Related Treatment-Emergent Adverse Events
Description: An AE was any untoward medical occurrence in a clinical investigation patient administered a study drug, regardless of causal attribution. TEAEs were defined as AEs with onset date on or after the first dose of study drug and no later than 30 days after the date of last study drug administration or start of a new study drug of anti-neoplasm therapy, whichever was earlier. Treatment related AEs were defined as AEs collected later than 30 days after the last study drug date or start of a new study drug of anti-neoplasm therapy.
Time Frame: From the first dose of study drug (Day 1) up to 30 days after the last dose of study drug, approximately 27 months
Population: The FAS included all patients who received at least 1 dose of HMPL-689.
Measure: Count of Participants; unit: Participants
Arm/Group | Dose Expansion Stage: CLL/SLL | Dose Expansion Stage: FL | Dose Expansion Stage: MZL | Dose Expansion Stage: LPL/WM | Dose Expansion Stage: MCL
Number analyzed (Participants) | 3 | 13 | 6 | 3 | 5
Participants
  Any TEAE | 3 | 13 | 5 | 3 | 5
  Any TRAE | 3 | 12 | 5 | 2 | 4

4. Secondary Outcome: Dose Escalation and Dose Expansion Stages: Objective Response Rate (ORR)
Description: ORR: percentage of patients with complete response (CR),CR with incomplete marrow recovery (CRi),nodular partial response (nPR),PR with lymphocytosis (PR-L) or PR for CLL patients; CR, very good PR (VGPR),PR or minor response (MR) for WM patients;CR or PR for patients with disease other than CLL and WM.CR: absence of serum (S) monoclonal immunoglobulin (Ig)M, normal S IgM, complete resolution of extramedullary disease,morphologically normal bone marrow aspirate and trephine biopsy. CRi:criteria fulfilled for CR but persistent cytopenia,anemia,thrombocytopenia or neutropenia. nPR:patients with residual CLL cells.PR-L:patients achieved PR with CLL-related signs/symptoms other than lymphocytosis and continued on therapy.PR, VGPR, MR: detectable monoclonal IgM,no new signs/symptoms of active disease and PR: ≥50% but <90% reduction in S IgM,reduction in extramedullary disease,VGPR: >=90% reduction in S IgM,complete resolution of extramedullary disease,MR: >=25% but <50% reduction in S IgM.
Time Frame: Tumor assessments performed every 8 weeks (+/-7 days) for the first 24 weeks and every 12 weeks (+/-7days) thereafter, up to a maximum of 58 months
Population: The efficacy analysis set (EAS) included all patients who received at least 1 dose of HMPL-689 and had a baseline tumor assessment and at least 1 evaluable post-baseline assessment unless death occurred before the first post-baseline assessment.
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | Dose Escalation Stage: HMPL-689 5 mg QD | Dose Escalation Stage: HMPL-689 10 mg QD | Dose Escalation Stage: HMPL-689 15 mg QD | Dose Escalation Stage: HMPL-689 20 mg QD | Dose Escalation Stage: HMPL-689 25 mg QD | Dose Escalation Stage: HMPL-689 30 mg QD | Dose Expansion Stage: CLL/SLL | Dose Expansion Stage: FL | Dose Expansion Stage: MZL | Dose Expansion Stage: LPL/WM | Dose Expansion Stage: MCL
Number analyzed (Participants) | 3 | 3 | 5 | 2 | 5 | 3 | 3 | 13 | 6 | 2 | 4
percentage of patients | 33.3 [0.8 to 90.6] | 66.7 [9.4 to 99.2] | 80.0 [28.4 to 99.5] | 100.0 [15.8 to 100.0] | 60.0 [14.7 to 94.7] | 66.7 [9.4 to 99.2] | 66.7 [9.4 to 99.2] | 84.6 [54.6 to 98.1] | 50.0 [11.8 to 88.2] | 100.0 [15.8 to 100.0] | 100.0 [39.8 to 100.0]

5. Secondary Outcome: Dose Escalation and Dose Expansion Stages: Time to Response (TTR)
Description: TTR was defined as the time from the first dose of study drug to the first occurrence of CR, CRi, PR, nPR, VGPR, PR-L, or MR. CR: absence of serum monoclonal IgM, normal serum IgM, complete resolution of extramedullary disease, morphologically normal bone marrow aspirate and trephine biopsy. CRi: criteria fulfilled for CR but persistent cytopenia, anemia, thrombocytopenia or neutropenia. PR: detectable monoclonal IgM, no new signs/symptoms of active disease, 50% but <90% reduction in serum IgM, reduction in extramedullary disease. nPR: patients with residual CLL cells. VGPR: detectable monoclonal IgM, no new signs/symptoms of active disease,>=90% reduction in serum IgM, complete resolution of extramedullary disease. PR-L: patients achieved PR with CLL-related signs/symptoms other than lymphocytosis and continued on therapy. MR: detectable monoclonal IgM, no new signs/symptoms of active disease, >=25% but <50% reduction in serum IgM.
Time Frame: as for outcome 4
Population: The EAS included all patients who received at least 1 dose of HMPL-689 and had a baseline tumor assessment and at least 1 evaluable post-baseline assessment unless death occurred before the first post-baseline assessment. Only patients with CR, CRi, PR, nPR, VGPR, PR-L, or MR were included in the analysis.
Measure: Median (Full Range); unit: months
Arm/Group | Dose Escalation Stage: HMPL-689 5 mg QD | Dose Escalation Stage: HMPL-689 10 mg QD | Dose Escalation Stage: HMPL-689 15 mg QD | Dose Escalation Stage: HMPL-689 20 mg QD | Dose Escalation Stage: HMPL-689 25 mg QD | Dose Escalation Stage: HMPL-689 30 mg QD | Dose Expansion Stage: CLL/SLL | Dose Expansion Stage: FL | Dose Expansion Stage: MZL | Dose Expansion Stage: LPL/WM | Dose Expansion Stage: MCL
Number analyzed (Participants) | 1 | 2 | 4 | 2 | 3 | 2 | 2 | 11 | 3 | 2 | 4
months | 1.87 [1.87 to 1.87] | 1.72 [1.68 to 1.77] | 8.80 [1.91 to 19.55] | 1.77 [1.68 to 1.87] | 2.27 [1.87 to 11.14] | 1.84 [1.84 to 1.84] | 2.81 [1.87 to 3.75] | 1.74 [1.64 to 2.07] | 2.53 [1.91 to 2.79] | 3.73 [1.84 to 5.62] | 1.76 [1.71 to 1.84]

6. Secondary Outcome: Dose Escalation and Dose Expansion Stages: Duration of Response (DOR)
Description: DOR: time from when first response (CR, CRi, PR, nPR, VGPR, PR-L and MR) was achieved until earlier of first documentation of definitive PD or death from any cause, whichever was earlier. CR: absence of S monoclonal IgM, normal S IgM, complete resolution of extramedullary disease, morphologically normal bone marrow aspirate and trephine biopsy. CRi: criteria fulfilled for CR but persistent cytopenia, anemia, thrombocytopenia or neutropenia. nPR: patients with residual CLL cells. PR-L: patients achieved PR with CLL-related signs/symptoms other than lymphocytosis and continued on therapy. PR, VGPR, MR: detectable monoclonal IgM, no new signs/symptoms of active disease and PR: ≥50% but <90% reduction in S IgM, reduction in extramedullary disease, VGPR: >=90% reduction in S IgM, complete resolution of extramedullary disease, MR: >=25% but <50% reduction in S IgM. PD: >=25% increase in S IgM level from lowest nadir and/or progression in clinical features attributable to the disease.
Time Frame: as for outcome 4
Population: as for outcome 5
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Dose Escalation Stage: HMPL-689 5 mg QD | Dose Escalation Stage: HMPL-689 10 mg QD | Dose Escalation Stage: HMPL-689 15 mg QD | Dose Escalation Stage: HMPL-689 20 mg QD | Dose Escalation Stage: HMPL-689 25 mg QD | Dose Escalation Stage: HMPL-689 30 mg QD | Dose Expansion Stage: CLL/SLL | Dose Expansion Stage: FL | Dose Expansion Stage: MZL | Dose Expansion Stage: LPL/WM | Dose Expansion Stage: MCL
Number analyzed (Participants) | 1 | 2 | 4 | 2 | 3 | 2 | 2 | 11 | 3 | 2 | 4
months | 1.9 [NA to NA] — NA indicates that upper and lower limits of confidence interval (CI) were not estimable due to insufficient number of patients with events at study closure. | 31.9 [NA to NA] — NA indicates that upper and lower limits of CI were not estimable due to insufficient number of patients with events at study closure. | 13.7 [12.6 to NA] — NA indicates that upper limit of CI was not estimable due to insufficient number of patients with events at study closure. | NA [9.3 to NA] — NA indicates that median and upper limit of CI were not estimable due to insufficient number of patients with events at study closure. | NA [NA to NA] — NA indicates that median, upper and lower limits of CI were not estimable due to insufficient number of patients with events at study closure. | NA [1.9 to NA] — NA indicates that median and upper limit of CI were not estimable due to insufficient number of patients with events at study closure. | NA [4.6 to NA] — NA indicates that median and upper limit of CI were not estimable due to insufficient number of patients with events at study closure. | NA [1.9 to NA] — NA indicates that median and upper limit of CI were not estimable due to insufficient number of patients with events at study closure. | NA [NA to NA] — NA indicates that median, upper and lower limits of CI were not estimable due to insufficient number of patients with events at study closure. | NA [4.9 to NA] — NA indicates that median and upper limit of CI were not estimable due to insufficient number of patients with events at study closure. | 9.1 [3.7 to NA] — NA indicates that upper limit of CI was not estimable due to insufficient number of patients with events at study closure.

7. Secondary Outcome: Dose Escalation and Dose Expansion Stages: Clinical Benefit Rate (CBR)
Description: CBR was defined as percentage of patients who had best overall response (BOR) with stable disease (SD) or better. BOR was defined as the best response recorded from the start of treatment until PD or new anti-cancer therapy, whichever came earlier. PD: >=25% increase in serum IgM level from lowest nadir and/or progression in clinical features attributable to the disease. SD: detectable monoclonal IgM, <25% reduction and <25% increase in serum IgM level, no progression in extramedullary disease, no new signs/symptoms of active disease.
Time Frame: Tumor assessments performed every 8 weeks (+/-7 days) for the first 24 weeks and every 12 weeks (+/-7 days) thereafter, up to a maximum of 58 months
Population: The EAS included all patients who received at least 1 dose of HMPL-689 and had a baseline tumor assessment and at least 1 evaluable post-baseline assessment unless death occurred before the first post-baseline assessment.
Measure: Number (95% Confidence Interval); unit: percentage of patients
Groups:
- Dose Escalation Stage: HMPL-689 10 mg QD: Patients received HMPL-689 10 mg QD orally for continuous 28-day treatment cycles until stage, death, intolerable toxicity, investigator's assessment of no benefit from the study treatment, withdrawal from the study, or the end of study, whichever occurred first.
Arm/Group | Dose Escalation Stage: HMPL-689 5 mg QD | Dose Escalation Stage: HMPL-689 10 mg QD | Dose Escalation Stage: HMPL-689 15 mg QD | Dose Escalation Stage: HMPL-689 20 mg QD | Dose Escalation Stage: HMPL-689 25 mg QD | Dose Escalation Stage: HMPL-689 30 mg QD | Dose Expansion Stage: CLL/SLL | Dose Expansion Stage: FL | Dose Expansion Stage: MZL | Dose Expansion Stage: LPL/WM | Dose Expansion Stage: MCL
Number analyzed (Participants) | 3 | 3 | 5 | 2 | 5 | 3 | 3 | 13 | 6 | 2 | 4
percentage of patients | 100.0 [29.2 to 100.0] | 100.0 [29.2 to 100.0] | 80.0 [28.4 to 99.5] | 100.0 [15.8 to 100.0] | 80.0 [28.4 to 99.5] | 66.7 [9.4 to 99.2] | 100.0 [29.2 to 100.0] | 84.6 [54.6 to 98.1] | 83.3 [35.9 to 99.6] | 100.0 [15.8 to 100.0] | 100.0 [39.8 to 100.0]

8. Secondary Outcome: Dose Escalation and Dose Expansion Stages: Progression-Free Survival (PFS)
Description: PFS was defined as the time from the date of first study drug to the earliest date of PD or death of any cause, whichever occurred first. PD was defined as >=25% increase in serum IgM level from lowest nadir and/or progression in clinical features attributable to the disease.
Time Frame: as for outcome 7
Population: The FAS included all patients who received at least 1 dose of HMPL-689.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Dose Escalation Stage: HMPL-689 5 mg QD | Dose Escalation Stage: HMPL-689 10 mg QD | Dose Escalation Stage: HMPL-689 15 mg QD | Dose Escalation Stage: HMPL-689 20 mg QD | Dose Escalation Stage: HMPL-689 25 mg QD | Dose Escalation Stage: HMPL-689 30 mg QD | Dose Expansion Stage: CLL/SLL | Dose Expansion Stage: FL | Dose Expansion Stage: MZL | Dose Expansion Stage: LPL/WM | Dose Expansion Stage: MCL
Number analyzed (Participants) | 3 | 3 | 5 | 3 | 6 | 3 | 3 | 13 | 6 | 3 | 5
months | 5.3 [3.8 to NA] — NA indicates that upper limit of CI was not estimable due to insufficient number of patients with events at study closure. | 33.6 [NA to NA] — NA indicates that upper and lower limits of CI were not estimable due to insufficient number of patients with events at study closure. | 16.6 [1.9 to NA] — NA indicates that upper limit of CI was not estimable due to insufficient number of patients with events at study closure. | NA [11.0 to NA] — NA indicates that median and upper limit of CI were not estimable due to insufficient number of patients with events at study closure. | 13.6 [1.8 to NA] — NA indicates that upper limit of CI was not estimable due to insufficient number of patients with events at study closure. | 3.7 [1.7 to NA] — NA indicates that upper limit of CI was not estimable due to insufficient number of patients with events at study closure. | NA [8.3 to NA] — NA indicates that median and upper limit of CI were not estimable due to insufficient number of patients with events at study closure. | 11.9 [1.8 to NA] — NA indicates that upper limit of CI was not estimable due to insufficient number of patients with events at study closure. | 5.6 [2.1 to NA] — NA indicates that upper limit of CI was not estimable due to insufficient number of patients with events at study closure. | NA [10.4 to NA] — NA indicates that median and upper limit of CI were not estimable due to insufficient number of patients with events at study closure. | 10.8 [5.5 to NA] — NA indicates that upper limit of CI was not estimable due to insufficient number of patients with events at study closure.

9. Secondary Outcome: Dose Escalation Stage: Plasma Concentration of HMPL-689
Description: Blood samples were collected to determine plasma concentration of HMPL-689. The pharmacokinetic (PK) parameters were determined by non-compartmental analysis.
Time Frame: Pre-dose on Days 1, 2, 15, 16, 28 of Cycle 1 and on Day 1 of Cycle 2; 0.5, 1, 2, 4 and 8 hours post-dose on Days 1, 15 and 28 of Cycle 1 (each cycle is 28 days)
Population: The pharmacokinetic analysis set (PKAS) included all patients who received at least 1 dose of HMPL-689 and had at least 1 PK sample obtained and analyzed. Only patients with data collected at specified timepoints are reported.
Measure: Mean (Standard Deviation); unit: nanograms per milliliter (ng/mL)
Arm/Group | Dose Escalation Stage: HMPL-689 5 mg QD | Dose Escalation Stage: HMPL-689 10 mg QD | Dose Escalation Stage: HMPL-689 15 mg QD | Dose Escalation Stage: HMPL-689 20 mg QD | Dose Escalation Stage: HMPL-689 25 mg QD | Dose Escalation Stage: HMPL-689 30 mg QD
Number analyzed (Participants) | 3 | 3 | 5 | 3 | 6 | 3
nanograms per milliliter (ng/mL)
  Pre-dose: Day 1 Cycle 1 | 0.000 (0.000) | 0.000 (0.000) | 0.000 (0.000) | 0.000 (0.000) | 0.000 (0.000) | 0.000 (0.000)
  0.5 hour post-dose: Day 1 Cycle 1: number analyzed (Participants) | 3 | 3 | 5 | 3 | 5 | 3
  0.5 hour post-dose: Day 1 Cycle 1 | 1.153 (1.220) | 65.133 (72.976) | 19.322 (18.574) | 87.733 (68.441) | 47.424 (78.327) | 36.907 (32.999)
  1 hour post-dose: Day 1 Cycle 1: number analyzed (Participants) | 3 | 3 | 5 | 3 | 5 | 3
  1 hour post-dose: Day 1 Cycle 1 | 14.457 (14.965) | 71.346 (63.493) | 66.740 (41.460) | 125.100 (78.083) | 110.780 (70.347) | 184.000 (176.952)
  2 hours post-dose: Day 1 Cycle 1 | 22.200 (4.629) | 50.887 (41.833) | 98.260 (16.955) | 108.067 (27.749) | 141.600 (82.032) | 167.033 (75.883)
  4 hours post-dose: Day 1 Cycle 1 | 19.267 (4.186) | 44.467 (22.299) | 95.260 (33.323) | 67.367 (30.596) | 103.700 (33.787) | 111.533 (49.843)
  8 hours post-dose: Day 1 Cycle 1: number analyzed (Participants) | 3 | 3 | 5 | 3 | 5 | 3
  8 hours post-dose: Day 1 Cycle 1 | 15.100 (4.190) | 35.867 (9.063) | 48.440 (18.373) | 36.700 (13.981) | 68.120 (27.164) | 72.600 (19.128)
  Pre-dose: Day 2 Cycle 1 | 4.490 (1.360) | 11.527 (6.411) | 12.442 (5.112) | 8.887 (4.148) | 20.017 (8.614) | 13.433 (1.501)
  Pre-dose: Day 15 Cycle 1: number analyzed (Participants) | 3 | 3 | 4 | 3 | 6 | 3
  Pre-dose: Day 15 Cycle 1 | 4.580 (0.521) | 35.613 (39.872) | 12.450 (9.931) | 11.100 (10.026) | 29.250 (14.562) | 22.900 (11.077)
  0.5 hour post-dose: Day 15 Cycle 1: number analyzed (Participants) | 3 | 3 | 4 | 3 | 5 | 3
  0.5 hour post-dose: Day 15 Cycle 1 | 5.443 (2.145) | 118.433 (82.709) | 44.295 (40.717) | 59.667 (52.905) | 45.180 (29.456) | 21.733 (9.166)
  1 hour post-dose: Day 15 Cycle 1: number analyzed (Participants) | 3 | 3 | 4 | 3 | 5 | 3
  1 hour post-dose: Day 15 Cycle 1 | 19.300 (26.414) | 115.400 (69.730) | 66.900 (50.101) | 100.667 (63.801) | 94.420 (72.734) | 116.667 (16.773)
  2 hours post-dose: Day 15 Cycle 1: number analyzed (Participants) | 3 | 3 | 4 | 3 | 5 | 3
  2 hours post-dose: Day 15 Cycle 1 | 31.123 (24.388) | 79.867 (23.500) | 86.425 (42.718) | 102.900 (22.999) | 122.220 (86.832) | 187.333 (88.636)
  4 hours post-dose: Day 15 Cycle 1: number analyzed (Participants) | 3 | 3 | 4 | 3 | 5 | 3
  4 hours post-dose: Day 15 Cycle 1 | 20.323 (11.020) | 56.200 (22.311) | 91.625 (31.814) | 97.667 (14.468) | 153.400 (30.345) | 158.833 (63.135)
  8 hours post-dose: Day 15 Cycle 1: number analyzed (Participants) | 3 | 3 | 3 | 2 | 5 | 3
  8 hours post-dose: Day 15 Cycle 1 | 15.933 (2.307) | 37.533 (16.861) | 73.233 (14.758) | 58.450 (9.122) | 87.620 (26.685) | 77.367 (25.143)
  Pre-dose: Day 16 Cycle 1: number analyzed (Participants) | 3 | 3 | 4 | 2 | 5 | 3
  Pre-dose: Day 16 Cycle 1 | 5.567 (0.958) | 61.367 (87.227) | 17.825 (4.234) | 15.100 (1.556) | 31.320 (13.989) | 20.267 (9.393)
  Pre-dose: Day 28 Cycle 1: number analyzed (Participants) | 3 | 2 | 4 | 3 | 5 | 3
  Pre-dose: Day 28 Cycle 1 | 5.837 (1.257) | 10.885 (1.860) | 19.575 (9.215) | 25.133 (7.251) | 32.380 (17.181) | 21.200 (10.121)
  0.5 hour post-dose: Day 28 Cycle 1: number analyzed (Participants) | 3 | 2 | 4 | 3 | 5 | 3
  0.5 hour post-dose: Day 28 Cycle 1 | 17.383 (22.271) | 101.100 (56.427) | 39.950 (37.487) | 67.000 (66.731) | 42.940 (18.447) | 24.367 (16.404)
  1 hour post-dose: Day 28 Cycle 1: number analyzed (Participants) | 3 | 2 | 4 | 3 | 5 | 3
  1 hour post-dose: Day 28 Cycle 1 | 24.473 (29.361) | 110.300 (46.245) | 56.150 (51.474) | 113.333 (85.096) | 101.740 (64.018) | 140.533 (137.107)
  2 hours post-dose: Day 28 Cycle 1: number analyzed (Participants) | 3 | 2 | 4 | 3 | 5 | 2
  2 hours post-dose: Day 28 Cycle 1 | 21.803 (15.134) | 61.550 (14.779) | 108.175 (39.401) | 126.500 (78.665) | 149.460 (74.134) | 219.250 (186.323)
  4 hours post-dose: Day 28 Cycle 1: number analyzed (Participants) | 3 | 2 | 4 | 3 | 5 | 3
  4 hours post-dose: Day 28 Cycle 1 | 25.767 (2.050) | 55.750 (22.698) | 111.950 (33.596) | 115.000 (22.068) | 145.720 (57.106) | 133.333 (17.559)
  8 hours post-dose: Day 28 Cycle 1: number analyzed (Participants) | 3 | 2 | 4 | 3 | 5 | 3
  8 hours post-dose: Day 28 Cycle 1 | 16.700 (3.341) | 32.700 (4.667) | 62.750 (21.418) | 66.867 (14.230) | 97.560 (29.737) | 81.533 (12.052)
  Pre-dose: Day 1 Cycle 2: number analyzed (Participants) | 3 | 2 | 5 | 2 | 5 | 3
  Pre-dose: Day 1 Cycle 2 | 8.593 (4.588) | 17.500 (7.292) | 17.880 (7.265) | 19.200 (2.121) | 30.400 (13.557) | 16.833 (5.341)

10. Secondary Outcome: Dose Escalation Stage: Plasma Trough Concentration (Ctrough) of HMPL-689
Description: Blood samples were collected to determine Ctrough of HMPL-689. The PK parameters were determined by non-compartmental analysis.
Time Frame: Days 1, 2, 15, 16, 28 of Cycle 1 and Day 1 of Cycle 2 (each cycle is 28 days)
Population: The PKAS included all patients who received at least 1 dose of HMPL-689 and had at least 1 PK sample obtained and analyzed. Only patients with data collected at specified timepoints are reported.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Dose Escalation Stage: HMPL-689 5 mg QD | Dose Escalation Stage: HMPL-689 10 mg QD | Dose Escalation Stage: HMPL-689 15 mg QD | Dose Escalation Stage: HMPL-689 20 mg QD | Dose Escalation Stage: HMPL-689 25 mg QD | Dose Escalation Stage: HMPL-689 30 mg QD
Number analyzed (Participants) | 3 | 3 | 5 | 3 | 6 | 3
ng/mL
  Day 1: Cycle 1: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0
  Day 2: Cycle 1: number analyzed (Participants) | 3 | 2 | 5 | 3 | 6 | 3
  Day 2: Cycle 1 | 4.490 (1.360) | 8.290 (4.398) | 12.442 (5.112) | 8.887 (4.148) | 20.017 (8.614) | 13.433 (1.501)
  Day 15: Cycle 1: number analyzed (Participants) | 3 | 3 | 3 | 2 | 5 | 3
  Day 15: Cycle 1 | 4.580 (0.521) | 35.613 (39.872) | 16.600 (6.678) | 16.650 (4.031) | 31.160 (15.418) | 22.900 (11.077)
  Day 16: Cycle 1: number analyzed (Participants) | 3 | 2 | 4 | 0 | 5 | 3
  Day 16: Cycle 1 | 5.567 (0.958) | 11.050 (5.162) | 17.825 (4.234) |  | 31.320 (13.989) | 20.267 (9.393)
  Day 28: Cycle 1: number analyzed (Participants) | 3 | 2 | 4 | 3 | 5 | 3
  Day 28: Cycle 1 | 5.837 (1.257) | 10.885 (1.860) | 19.575 (9.215) | 25.133 (7.251) | 32.380 (17.181) | 21.200 (10.121)
  Day 1: Cycle 2: number analyzed (Participants) | 2 | 3 | 5 | 2 | 5 | 3
  Day 1: Cycle 2 | 6.140 (2.447) | 17.500 (7.292) | 17.880 (7.265) | 19.200 (2.121) | 30.400 (13.557) | 16.833 (5.341)

11. Secondary Outcome: Dose Expansion Stage: Plasma Concentration of HMPL-689
Description: Blood samples were collected to determine plasma concentration of HMPL-689. The PK parameters were determined by non-compartmental analysis.
Time Frame: Pre-dose on Day 1 of Cycles 1, 2, 3, 5, 7, 9, 11, 13 and on Day 15 of Cycle 1; 0 hour on Day 1 of Cycle 1; 1, 2, 3, 4 hours post-dose on Days 1 and 15 of Cycle 1 (each cycle is 28 days)
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Dose Expansion Stage: CLL/SLL | Dose Expansion Stage: FL | Dose Expansion Stage: MZL | Dose Expansion Stage: LPL/WM | Dose Expansion Stage: MCL
Number analyzed (Participants) | 3 | 13 | 6 | 3 | 5
ng/mL
  Pre-dose: Day 1 Cycle 1 | 0.000 (0.000) | 1.685 (6.074) | 0.000 (0.000) | 0.000 (0.000) | 0.000 (0.000)
  0 hour post-dose: Day 1 Cycle 1: number analyzed (Participants) | 0 | 3 | 0 | 0 | 1
  0 hour post-dose: Day 1 Cycle 1 |  | 48.400 (61.060) |  |  | NA (NA) — NA indicates that mean and standard deviation (SD) were not estimable for n<3, as pre-specified in the statistical analysis plan (SAP).
  1 hour post-dose: Day 1 Cycle 1: number analyzed (Participants) | 3 | 12 | 6 | 3 | 4
  1 hour post-dose: Day 1 Cycle 1 | 54.743 (85.161) | 108.857 (74.766) | 145.600 (131.539) | 86.950 (93.589) | 75.750 (33.441)
  2 hours post-dose: Day 1 Cycle 1 | 104.233 (117.306) | 150.523 (51.261) | 171.000 (71.632) | 136.333 (114.031) | 132.460 (27.338)
  3 hours post-dose: Day 1 Cycle 1: number analyzed (Participants) | 3 | 12 | 6 | 3 | 3
  3 hours post-dose: Day 1 Cycle 1 | 101.967 (70.324) | 130.742 (54.780) | 131.600 (33.368) | 98.267 (70.926) | 116.667 (11.930)
  4 hours post-dose: Day 1 Cycle 1 | 111.833 (22.661) | 117.708 (62.408) | 108.833 (30.521) | 72.933 (37.302) | 119.720 (36.898)
  Pre-dose: Day 15 Cycle 1: number analyzed (Participants) | 3 | 12 | 6 | 3 | 5
  Pre-dose: Day 15 Cycle 1 | 22.933 (8.804) | 37.056 (22.923) | 31.363 (25.923) | 16.667 (16.220) | 115.880 (147.709)
  1 hour post-dose: Day 15 Cycle 1: number analyzed (Participants) | 3 | 12 | 6 | 3 | 5
  1 hour post-dose: Day 15 Cycle 1 | 142.967 (119.865) | 146.358 (92.001) | 125.917 (52.229) | 95.467 (66.718) | 180.800 (87.697)
  2 hours post-dose: Day 15 Cycle 1: number analyzed (Participants) | 3 | 12 | 6 | 3 | 5
  2 hours post-dose: Day 15 Cycle 1 | 233.667 (2.082) | 193.417 (92.573) | 167.433 (71.148) | 128.000 (88.705) | 190.400 (53.003)
  3 hours post-dose: Day 15 Cycle 1: number analyzed (Participants) | 3 | 12 | 6 | 3 | 4
  3 hours post-dose: Day 15 Cycle 1 | 179.000 (30.447) | 166.550 (65.746) | 140.867 (56.317) | 95.333 (38.783) | 165.000 (75.024)
  4 hours post-dose: Day 15 Cycle 1: number analyzed (Participants) | 3 | 12 | 6 | 3 | 5
  4 hours post-dose: Day 15 Cycle 1 | 140.667 (48.003) | 148.333 (44.252) | 123.483 (48.346) | 85.167 (35.335) | 153.520 (46.202)
  Pre-dose: Day 1 Cycle 2: number analyzed (Participants) | 2 | 12 | 5 | 3 | 5
  Pre-dose: Day 1 Cycle 2 | NA (NA) — NA indicates that mean and SD were not estimable for n<3, as pre-specified in the SAP. | 61.493 (69.318) | 30.666 (23.182) | 15.237 (5.614) | 37.060 (25.195)
  Pre-dose: Day 1 Cycle 3: number analyzed (Participants) | 3 | 9 | 4 | 3 | 4
  Pre-dose: Day 1 Cycle 3 | 32.633 (15.667) | 39.367 (36.625) | 41.815 (34.757) | 12.890 (8.707) | 43.800 (13.444)
  Pre-dose: Day 1 Cycle 5: number analyzed (Participants) | 2 | 5 | 5 | 2 | 3
  Pre-dose: Day 1 Cycle 5 | NA (NA) — NA indicates that mean and SD were not estimable for n<3, as pre-specified in the SAP. | 82.100 (55.917) | 40.412 (40.658) | NA (NA) — NA indicates that mean and SD were not estimable for n<3, as pre-specified in the SAP. | 25.167 (25.877)
  Pre-dose: Day 1 Cycle 7: number analyzed (Participants) | 2 | 2 | 3 | 3 | 3
  Pre-dose: Day 1 Cycle 7 | NA (NA) — NA indicates that mean and SD were not estimable for n<3, as pre-specified in the SAP. | NA (NA) — NA indicates that mean and SD were not estimable for n<3, as pre-specified in the SAP. | 23.983 (35.772) | 19.733 (11.057) | 75.967 (54.444)
  Pre-dose: Day 1 Cycle 9: number analyzed (Participants) | 1 | 3 | 1 | 3 | 2
  Pre-dose: Day 1 Cycle 9 | NA (NA) — NA indicates that mean and SD were not estimable for n<3, as pre-specified in the SAP. | 49.400 (46.088) | NA (NA) — NA indicates that mean and SD were not estimable for n<3, as pre-specified in the SAP. | 18.533 (10.883) | NA (NA) — NA indicates that mean and SD were not estimable for n<3, as pre-specified in the SAP.
  Pre-dose: Day 1 Cycle 11: number analyzed (Participants) | 1 | 2 | 1 | 2 | 0
  Pre-dose: Day 1 Cycle 11 | NA (NA) — NA indicates that mean and SD were not estimable for n<3, as pre-specified in the SAP. | NA (NA) — NA indicates that mean and SD were not estimable for n<3, as pre-specified in the SAP. | NA (NA) — NA indicates that mean and SD were not estimable for n<3, as pre-specified in the SAP. | NA (NA) — NA indicates that mean and SD were not estimable for n<3, as pre-specified in the SAP. |
  Pre-dose: Day 1 Cycle 13: number analyzed (Participants) | 0 | 1 | 1 | 1 | 0
  Pre-dose: Day 1 Cycle 13 |  | NA (NA) — NA indicates that mean and SD were not estimable for n<3, as pre-specified in the SAP. | NA (NA) — NA indicates that mean and SD were not estimable for n<3, as pre-specified in the SAP. | NA (NA) — NA indicates that mean and SD were not estimable for n<3, as pre-specified in the SAP. |

12. Secondary Outcome: Dose Expansion Stage: Plasma Trough Concentration of HMPL-689
Description: as for outcome 10
Time Frame: Day 1 of Cycles 1, 2, 3, 5, 7, 9, 11, 13 and on Day 15 of Cycle 1 (each cycle is 28 days)
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Dose Expansion Stage: CLL/SLL | Dose Expansion Stage: FL | Dose Expansion Stage: MZL | Dose Expansion Stage: LPL/WM | Dose Expansion Stage: MCL
Number analyzed (Participants) | 3 | 12 | 6 | 3 | 4
ng/mL
  Day 1: Cycle 1: number analyzed (Participants) | 0 | 1 | 0 | 0 | 0
  Day 1: Cycle 1 |  | 21.900 (NA) — NA indicates that SD could not be determined when only 1 patient was analyzed. |  |  |
  Day 15: Cycle 1 | 22.933 (8.804) | 37.056 (22.923) | 31.363 (25.923) | 16.667 (16.220) | 132.125 (165.321)
  Day 1: Cycle 2: number analyzed (Participants) | 2 | 9 | 5 | 3 | 4
  Day 1: Cycle 2 | 24.550 (2.758) | 41.013 (36.989) | 30.666 (23.182) | 15.237 (5.614) | 46.325 (16.555)
  Day 1: Cycle 3: number analyzed (Participants) | 2 | 7 | 3 | 2 | 4
  Day 1: Cycle 3 | 23.750 (4.172) | 46.214 (38.254) | 33.587 (37.495) | 14.390 (11.752) | 43.800 (13.444)
  Day 1: Cycle 5: number analyzed (Participants) | 2 | 4 | 4 | 2 | 3
  Day 1: Cycle 5 | 36.450 (15.627) | 63.625 (43.513) | 49.225 (41.065) | 18.150 (11.102) | 25.167 (25.877)
  Day 1: Cycle 7: number analyzed (Participants) | 2 | 2 | 2 | 2 | 3
  Day 1: Cycle 7 | 34.050 (6.293) | 27.950 (9.829) | 32.550 (46.033) | 22.850 (13.647) | 75.967 (54.444)
  Day 1: Cycle 9: number analyzed (Participants) | 1 | 2 | 1 | 3 | 2
  Day 1: Cycle 9 | 37.400 (NA) — NA indicates that SD could not be determined when only 1 patient was analyzed. | 59.050 (60.740) | 61.600 (NA) — NA indicates that SD could not be determined when only 1 patient was analyzed. | 18.533 (10.883) | 28.950 (4.596)
  Day 1: Cycle 11: number analyzed (Participants) | 1 | 1 | 1 | 2 | 0
  Day 1: Cycle 11 | 28.100 (NA) — NA indicates that SD could not be determined when only 1 patient was analyzed. | 24.100 (NA) — NA indicates that SD could not be determined when only 1 patient was analyzed. | 65.200 (NA) — NA indicates that SD could not be determined when only 1 patient was analyzed. | 35.050 (30.193) |
  Day 1: Cycle 13: number analyzed (Participants) | 0 | 1 | 1 | 1 | 0
  Day 1: Cycle 13 |  | 29.600 (NA) — NA indicates that SD could not be determined when only 1 patient was analyzed. | 18.800 (NA) — NA indicates that SD could not be determined when only 1 patient was analyzed. | 17.300 (NA) — NA indicates that SD could not be determined when only 1 patient was analyzed. |

13. Secondary Outcome: Dose Escalation and Dose Expansion Stages: Change From Baseline in Corrected QT Interval (QTc) Using Fridericia Formula (QTcF)
Description: 12-lead electrocardiogram was performed to evaluate the effect of HMPL-689 on cardiac repolarization by detecting the changes in QTcF intervals. Baseline was defined as the last assessment performed prior to or on first non-zero dose date with time point marked as "pre-dose".
Time Frame: 2 and 4 hours on Baseline (Day 1) of Cycle 1; 0, 2 and 4 hours on Day 15 of Cycle 1 (dose escalation phase); 1, 2, 3 and 4 hours on Baseline (Day 1) of Cycle 1; 0, 1, 2, 3, and 4 hours on Day 15 of Cycle 1 (dose expansion phase) (each cycle is 28 days)
Population: The FAS included all patients who received at least 1 dose of HMPL-689. As pre-specified in the protocol, the results are presented by dose level and combined data for dose expansion stage is presented for all patients evaluable for this endpoint who received HMPL-689 at RP2D (30 mg QD) in dose expansion stage. Only patients with data collected at specified timepoints are reported.
Measure: Mean (Standard Deviation); unit: millisecond (msec)
Groups:
- Dose Expansion Stage: CLL/SLL, FL, MZL, LPL/WM, MCL: Patients with CLL/SLL, FL, MZL, LPL/WM, MCL received HMPL-689 at RP2D, that is, 30 mg QD orally for continuous 28-day treatment cycles until PD, death, intolerable toxicity, investigator's assessment of no benefit from the study treatment, withdrawal from the study, or the end of study, whichever occurred first.
Arm/Group | Dose Escalation Stage: HMPL-689 5 mg QD | Dose Escalation Stage: HMPL-689 10 mg QD | Dose Escalation Stage: HMPL-689 15 mg QD | Dose Escalation Stage: HMPL-689 20 mg QD | Dose Escalation Stage: HMPL-689 25 mg QD | Dose Escalation Stage: HMPL-689 30 mg QD | Dose Expansion Stage: CLL/SLL, FL, MZL, LPL/WM, MCL
Number analyzed (Participants) | 3 | 3 | 5 | 3 | 6 | 3 | 30
millisecond (msec)
  1 hour: Day 1 Cycle 1: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 30
  1 hour: Day 1 Cycle 1 |  |  |  |  |  |  | -5.14 (10.6)
  2 hours: Day 1 Cycle 1 | -6.89 (5.68) | 17.3 (0.471) | -10.4 (7.51) | -11.5 (9.19) | -13.3 (13.5) | -18.5 (2.59) | -1.43 (9.80)
  3 hours: Day 1 Cycle 1: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 30
  3 hours: Day 1 Cycle 1 |  |  |  |  |  |  | -2.21 (9.98)
  4 hours: Day 1 Cycle 1 | -8.33 (7.00) | 9.67 (5.66) | 2.27 (13.6) | 6.11 (5.82) | -9.33 (17.9) | -10.7 (8.82) | -2.46 (10.2)
  0 hour: Day 15 Cycle 1 | -11.3 (21.7) | -0.333 (8.49) | -2.17 (8.72) | -9.83 (2.59) | -4.33 (13.6) | -3.50 (4.01) | 0.231 (11.9)
  1 hour: Day 15 Cycle 1: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 30
  1 hour: Day 15 Cycle 1 |  |  |  |  |  |  | 2.11 (11.2)
  2 hours: Day 15 Cycle 1 | -10.6 (7.70) | 1.50 (3.06) | -0.583 (5.65) | -7.22 (7.83) | -10.0 (16.4) | -14.8 (10.6) | -0.524 (9.83)
  3 hours: Day 15 Cycle 1: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 30
  3 hours: Day 15 Cycle 1 |  |  |  |  |  |  | 0.614 (8.47)
  4 hours: Day 15 Cycle 1 | -13.1 (12.1) | 6.67 (12.7) | -2.17 (7.33) | -9.11 (10.9) | -4.27 (18.8) | -11.0 (11.7) | -0.964 (11.2)

ADVERSE EVENTS:
Time Frame: AEs and SAEs were collected from the first dose of study drug (Day 1) up to 30 days after the last dose of study drug, approximately 34 months for dose escalation stage and 27 months for dose expansion stage. All-cause mortality (deaths) were collected from the first dose of study drug (Day 1) up to 58 months.
Description: Analysis was performed on the FAS.
Arm/Group | Dose Escalation Stage: HMPL-689 5 mg QD | Dose Escalation Stage: HMPL-689 10 mg QD | Dose Escalation Stage: HMPL-689 15 mg QD | Dose Escalation Stage: HMPL-689 20 mg QD | Dose Escalation Stage: HMPL-689 25 mg QD | Dose Escalation Stage: HMPL-689 30 mg QD | Dose Expansion Stage: CLL/SLL | Dose Expansion Stage: FL | Dose Expansion Stage: MZL | Dose Expansion Stage: LPL/WM | Dose Expansion Stage: MCL
All-Cause Mortality (participants affected / at risk) | 0/3 | 1/3 | 1/5 | 0/3 | 0/6 | 0/3 | 0/3 | 0/13 | 0/6 | 1/3 | 2/5
Serious Adverse Events (participants affected / at risk) | 0/3 | 2/3 | 2/5 | 3/3 | 2/6 | 1/3 | 1/3 | 5/13 | 2/6 | 0/3 | 3/5
Other Adverse Events (participants affected / at risk) | 3/3 | 3/3 | 5/5 | 3/3 | 6/6 | 3/3 | 3/3 | 13/13 | 5/6 | 3/3 | 5/5
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dose Escalation Stage: HMPL-689 5 mg QD (N=3) | Dose Escalation Stage: HMPL-689 10 mg QD (N=3) | Dose Escalation Stage: HMPL-689 15 mg QD (N=5) | Dose Escalation Stage: HMPL-689 20 mg QD (N=3) | Dose Escalation Stage: HMPL-689 25 mg QD (N=6) | Dose Escalation Stage: HMPL-689 30 mg QD (N=3) | Dose Expansion Stage: CLL/SLL (N=3) | Dose Expansion Stage: FL (N=13) | Dose Expansion Stage: MZL (N=6) | Dose Expansion Stage: LPL/WM (N=3) | Dose Expansion Stage: MCL (N=5)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
COVID-19 (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Clostridium difficile colitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cytomegalovirus infection reactivation (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
COVID-19 pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pneumocystis jirovecii pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pyelonephritis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Colitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Colitis ulcerative (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Asthenia (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Disease progression (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Multiple fractures (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Epilepsy (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Psychotic disorder (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cutaneous vasculitis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Failure to thrive (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypercalcaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Renal failure (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dose Escalation Stage: HMPL-689 5 mg QD (N=3) | Dose Escalation Stage: HMPL-689 10 mg QD (N=3) | Dose Escalation Stage: HMPL-689 15 mg QD (N=5) | Dose Escalation Stage: HMPL-689 20 mg QD (N=3) | Dose Escalation Stage: HMPL-689 25 mg QD (N=6) | Dose Escalation Stage: HMPL-689 30 mg QD (N=3) | Dose Expansion Stage: CLL/SLL (N=3) | Dose Expansion Stage: FL (N=13) | Dose Expansion Stage: MZL (N=6) | Dose Expansion Stage: LPL/WM (N=3) | Dose Expansion Stage: MCL (N=5)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 1 (3) | 3 (10) | 1 (1) | 2 (2) | 0 (0) | 1 (4) | 5 (6) | 2 (2) | 1 (2) | 1 (3)
Haemorrhoids (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (5) | 0 (0) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 2 (3) | 0 (0) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (2) | 1 (1) | 0 (0) | 0 (0)
Gastrointestinal disorder (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haematemesis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Stomatitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 2 (3) | 0 (0) | 0 (0)
Swollen tongue (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Abdominal tenderness (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Anal rash (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Colitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Flatulence (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Lip swelling (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Melaena (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Odynophagia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Oral disorder (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Saliva altered (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
COVID-19 (Infections and infestations) | 0 (0) | 1 (2) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 4 (4) | 0 (0) | 1 (1) | 2 (2)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (5) | 2 (2) | 1 (2) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (4) | 1 (1) | 3 (7) | 1 (1) | 0 (0) | 0 (0)
Bronchitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Gastroenteritis viral (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lyme disease (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Onychomycosis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Subcutaneous abscess (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diarrhoea infectious (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Escherichia infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Escherichia urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Genital herpes simplex (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gingivitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Rash pustular (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tinea infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cutaneous vasculitis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 1 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (2) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2)
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 3 (4) | 0 (0) | 0 (0) | 0 (0)
Rash pruritic (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Skin lesion (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Night sweats (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 1 (1)
Eczema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Onychomadesis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Photosensitivity reaction (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin burning sensation (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Skin hypopigmentation (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 3 (3) | 1 (1) | 0 (0) | 2 (2)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 1 (3) | 1 (1) | 5 (6) | 1 (1) | 1 (2) | 0 (0)
Eosinophilia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Lymphadenopathy (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Neutrophilia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 1 (2) | 1 (1)
Blood alkaline phosphatase increased (Investigations) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 2 (3) | 0 (0) | 0 (0) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (2) | 1 (1)
Blood creatinine increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (3) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 2 (2)
Blood creatine phosphokinase increased (Investigations) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Electrocardiogram QT prolonged (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Platelet count decreased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
White blood cell count decreased (Investigations) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
White blood cell count increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lipase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 1 (2) | 0 (0)
Blood bilirubin increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Blood lactate dehydrogenase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (2)
Activated partial thromboplastin time prolonged (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Amylase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Blood cholesterol increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
CD4 lymphocytes decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
International normalised ratio increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Liver function test increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lymphocyte count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 0 (0)
Neutrophil count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Transaminases increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 1 (1) | 0 (0) | 4 (5) | 0 (0) | 0 (0) | 0 (0)
Bone pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (4) | 1 (1) | 0 (0) | 0 (0)
Spinal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 3 (4) | 1 (1) | 0 (0) | 1 (1)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Increased upper airway secretion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Respiratory tract inflammation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Bronchostenosis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Laryngeal haemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 1 (3) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 3 (3) | 1 (1) | 0 (0) | 0 (0)
Balance disorder (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Burning sensation (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Disturbance in attention (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1)
Hypoaesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Memory impairment (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dysgeusia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Paraesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Presyncope (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Fatigue (General disorders) | 0 (0) | 0 (0) | 1 (2) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 4 (4) | 0 (0) | 1 (1) | 2 (2)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 3 (3) | 2 (4) | 1 (2) | 1 (2)
Asthenia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Oedema peripheral (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vaccination site pain (General disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
General physical health deterioration (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Chills (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Facial pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Influenza like illness (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Malaise (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Mass (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Non-cardiac chest pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Peripheral swelling (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Dyslipidaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypocalcaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (4) | 0 (0) | 0 (0) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 3 (5) | 0 (0) | 0 (0) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (2) | 0 (0) | 1 (1)
Hyperuricaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hyperkalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypermagnesaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypophosphataemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Flushing (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Lymphoedema (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Phlebitis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Procedural pain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Angina pectoris (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bradycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Coronary artery disease (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Extrasystoles (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Periorbital oedema (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Retinopathy (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dry eye (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Erythema of eyelid (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Eye pruritus (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vision blurred (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Jarisch-Herxheimer reaction (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Seasonal allergy (Immune system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Middle ear inflammation (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Insomnia (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Anxiety (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Chronic kidney disease (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dysuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Leukocyturia (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Micturition urgency (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Urinary incontinence (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Colorectal adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Prostatitis (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)

LIMITATIONS AND CAVEATS:
The study was terminated based on strategic evaluation of the clinical development of HMPL-689 in the United States, Europe, and Australia with no safety concerns.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2022-12-12): https://cdn.clinicaltrials.gov/large-docs/26/NCT03786926/Prot_000.pdf
  • Statistical Analysis Plan (2024-07-22): https://cdn.clinicaltrials.gov/large-docs/26/NCT03786926/SAP_001.pdf